CLINICAL TRIAL: NCT01387659
Title: Study to Evaluate Tolerability of Myfortic With Simulect Induction and Tacrolimus Without Steroids in Three Patient Populations; 1: Kidney/Pancreas Transplants,2: Diabetic Kidney Transplants, and 3: Non-diabetic Kidney Transplants
Brief Title: Evaluate Tolerability of Myfortic®/Simulect® and Tacrolimus Without Steroids in Three Patient Populations
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to slow enrollment
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10-244
Record Dates: First submitted 2011-06-08; First posted 2011-07-04 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2013-09

CONDITIONS: Diabetes; Immunosuppression
Keywords: Myfortic; Simulect; Steroids; Diabetes; Transplant; Gastric emptying; Gastric motility
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Myfortic®/Simulect® and Tacrolimus Without Steroids in Three Patient Populations
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transplant recipients (Experimental): All subjects receive identical drug treatment
  Interventions: Procedure: Gastric emptying test

INTERVENTIONS:
Procedure: Gastric emptying test — Gastric emptying tests will be performed at baseline, 6 months and 12 months
  Other Names: Gastric motility

SUMMARY:
This study is designed to evaluate the tolerability of Myfortic®/Simulect® combination in diabetic patients in a steroid free regimen. Due to the diverse ethnicity of our transplant recipient population, the study will determine any different responses, including autoimmunity, between Hispanic, and Caucasian, patients.

DETAILED DESCRIPTION:
Myfortic® is an enteric-coated formulation of the sodium salt derivative of mycophenolic acid (MPA) that is administered to control kidney graft rejection. Myfortic® was developed to improve MPA-related upper gastrointestinal (GI) side effects by delaying the release of MPA until it reaches the large surface of the small bowel. Approximately half of all the kidney transplant recipients in the United States have diabetes mellitus. A recent analysis of approximately 30,000 kidney transplant recipients included in the U.S. Renal Data System showed that 42% of patients had pre-transplant diabetes (1). Moreover, 15% to 20% of patients develop diabetes after transplantation, a condition that is commonly known as post-diabetes mellitus (1-3). It was previously shown that the rate and extent of MPA absorption is minimally affected by diabetes (4). Limited data is available in the current literature on Myfortic® and Simulect® based therapy in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (age 18 to 65 years of age), male or female Hispanic or Caucasian.
2. Primary kidney or kidney transplant patients (cadaveric, living related, or living unrelated)
3. Written inform consent obtained. The patients are willing to participate in the study at UTMB.
4. Female with negative pregnancy test.
5. PRA < 20 %.
6. En-blocks and two kidneys (tx'd at the same time) will be allowed.
7. Cold Ischemia time ≤ 30 hrs
8. Hep C patients will be allowed to enroll in this study

Exclusion Criteria:

1. Multi-organ transplants
2. Transplant from non-heart beating donor (NHBD) or dual transplants
3. A-B-O incompatible or positive cross match
4. Conditions which significantly alter the absorption, distribution, and metabolism (except for diarrhea) of medications.
5. Women of childbearing potential not using contraception method(s) as well as women who are breastfeeding
6. Inability to tolerate oral medications
7. Inability to sign a written consent form or to cooperate with investigators
8. Use of an investigational medication in the past 30 days.
9. Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study (specify as required)
10. HIV positive patients
11. History of psychosocial instability
12. Mental incompetence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Tolerability of Myfortic in combination with Simulect and Tacrolimus without steroids | 24 months
  Assure that immunosuppression protects graft function by decreased incidence of rejection and side effects

SECONDARY OUTCOMES:
GI complications | 24 months
  Gastric emptying test
Graft function | 24 months
  Renal function assessed by serum creatinine and calculating creatinine clearance.
  Pancreas function assessed by glucose control, exogenous insulin requirement, HgbA1C
Biopsy proven rejection | 24 months
  Renal graft core biopsy will be performed on all suspected rejection.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Cicalese, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States